CLINICAL TRIAL: NCT01385072
Title: Pilot Study of Hematopoietic Stem Cell Transplantation From Two Matched Sibling Donors in Treating Patients With Poor Prognosis Acute Leukemia and Advanced Lymphoproliferative Malignancies
Status: Unknown | Phase: Phase 1 / Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Rabin Medical Center (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 6188
Record Dates: First submitted 2011-06-28; First posted 2011-06-29 (Estimated); Last update posted 2011-11-16 (Estimated); Status verified 2011-06

CONDITIONS: Relapsed and Refractory Acute Leukemia
Keywords: acute leukemia; relapse; induction failure; allogeneic transplantation; graft versus leukemia effect
MeSH Terms: conditions — Recurrence

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Double matched sibling transplantation (Experimental): Patients with poor risk active acute leukemia and who have 2 matched sibling donors can be included. Patients' conditioning may be myeloablative or non-myeloablative. Both matched donors will be mobilized with G-CSF and their peripheral blood stem cells will be collected on day 0.Equal numbers of CD34+ cells from both donors will be transfused to the patient.
  Patients will be followed for engraftment kinetics, chimerism, GVHD rate, severity and response to treatment, relapse rates, DFS and OS.
  Interventions: Biological: Double matched sibling transplantation

INTERVENTIONS:
Biological: Double matched sibling transplantation — Patients with poor risk active acute leukemia and who have 2 matched sibling donors can be included. Patients' conditioning may be myeloablative or non-myeloablative. Both matched donors will be mobilized with G-CSF and their peripheral blood stem cells will be collected on day 0.Equal numbers of CD34+ cells from both donors will be transfused to the patient.
  Patients will be followed for engraftment kinetics, chimerism, GVHD rate, severity and response to treatment, relapse rates, DFS and OS.

SUMMARY:
Patients with active acute leukemia have dismal prognoses even with allogeneic transplantation.Thus,new measures to enhance graft versus leukemia effect and reduce relapse rates are needed.

Relapse risk after double umbilical cord transplantations have been shown to be significantly lower compared to matched sibling and matched unrelated donor transplantations due to better graft versus leukemia effect.

The investigators hypothesize, that concomitant transplantation from 2 matched siblings may improve GVL effect and reduce relapse rate in patients with high risk acute leukemias and other high risk hematological malignancies.

ELIGIBILITY:
Inclusion Criteria:

1. Age 18 years or older
2. Patients with refractory or relapsed acute leukemia unable to receive myeloablative conditioning.
3. Patients with refractory or relapsed acute leukemia able to receive myeloablative conditioning but with the following factors:

   AML- 2 or more of the following: duration of CR1 < 6 months, poor cytogenetics, circulating blasts, karnofsky < 90.

   ALL- age > 40 or second and additional relapse, or 2 or more of the following: BM blasts > 25%, age 18-39,first refractory relapse, donor CMV positive.
4. Patients with 2 matched siblings and donor age > 18 years old.
5. Patients with advanced multiple myeloma with life expectancy of less than 6 months with standard therapy or transplantation.
6. Patients with advanced lymphoma with life expectancy of less than 6 months with standard therapy or transplantation.

Exclusion Criteria:

1. Patient age < 18 years.
2. Donor age < 18 years.
3. Patients in remission or not fulfilling above disease criteria -

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Estimated)
Dates: Start 2011-08; Primary Completion 2014-08 (Estimated); Study Completion 2015-04 (Estimated)

PRIMARY OUTCOMES:
Acute graft versus host disease rate,severity and response to treatment | 100 days

SECONDARY OUTCOMES:
relapse rate | 12 months

CONTACTS AND LOCATIONS:
Overall Officials: Moshe Yeshurun, MD, Principal Investigator — Davidoff cancer center, Beilinson hospital, Rabin Medical Center
Locations (1):
- Davidoff Cancer Center, Beilin hospital, Rabin medical center, Petah Tikva, Israel